CLINICAL TRIAL: NCT02957539
Title: Financial vs. Non-Financial Rewards for Weight Loss and Weight Maintenance: A Randomized Controlled Trial
Brief Title: Financial vs. Non-Financial Rewards for Weight Loss and Weight Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIR 15-459
Record Dates: First submitted 2016-11-01; First posted 2016-11-07 (Estimated); Results first posted 2023-03-31 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Obesity
Keywords: motivation; patient incentives
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- No Reward (No Intervention): At enrollment, participants randomized to usual care will be given the MOVE! workbook that serves both as an information resource on diet and exercise, a resource for tools to achieve weight loss goals, and a log of participants' goals, motivations, and outcomes. Each participant will be given a chart with a personalized target weight for a loss of 1lb. per week for 16 weeks. Participants will be given a digital scale or wireless scale and counseled to weigh themselves daily. Participants will enter their weight weekly into an online portal. They will also complete the surveys in the portal. They will receive text message reminders to enter their weight.
- Financial Reward Arm (Experimental): Same as usual care, plus financial rewards that are earned in two ways: an assured and random. For the assured reward, they will receive compensation at the end of each month that they are at or below their target weight on the last day of that period. For the random portion, each week that a participant is at or below their target weight, the patient is entered in random drawing to win additional compensation. Over the first eight weeks the patient has a 1-in-8 chance of winning.Over the 17-32 week period, Veterans in this group will receive token rewards for tracking and reporting their weekly weights regardless of whether it was on target. Each week that the patient enters his/her weight into the portal, he will have a 1-in-8 chance to earn the token reward, such as a t-shirt or movie tickets. Participants will enter their weight weekly into an online portal. They will also complete the surveys in the portal. They will receive text message reminders to enter their weight.
  Interventions: Behavioral: Financial rewards
- Non-financial Reward Arm (Experimental): Procedures for the non-financial rewards arm is identical to procedures for the financial reward arm, except that the Veteran will earn points rather than cash. Each week a random drawing will be for 20 points, each monthly weigh in is worth 5 points. Veterans will be given non-financial rewards associated with the number of points they earn.
  Interventions: Behavioral: Non-Financial rewards

INTERVENTIONS:
Behavioral: Financial rewards — Veterans in the financial reward arm receive all of the services of the usual care arm, plus rewards that are earned in two ways: an assured portion, and a random portion. For the assured reward, they will receive compensation at the end of each month (defined as a four week period) that they are at or below their target weight. For the random portion, each week that a participant is at or below their target weight, the patient is entered into a drawing to win additional compensation. Over the first eight weeks the patient has a 1-in-8 chance of winning. Over the 17-32 week period, Veterans in this group will receive token incentives for tracking and reporting their weekly weights regardless of whether it was on target. Each week that the patient enters their weight into the portal, s/he will have a 1-in-8 chance to earn the token incentive, such as a t-shirt or movie ticket. The participant will receive reminder text messages.
  Arms: Financial Reward Arm
Behavioral: Non-Financial rewards — Procedures for the non-financial rewards arm are identical to procedures for the financial reward arm, except that the Veteran will earn points rather than cash. Each weekly random drawing will be for 20 points. Veterans will choose non-financial rewards associated with the number of points they earn.
  Arms: Non-financial Reward Arm

SUMMARY:
Three of every four Veterans are overweight or obese, and weight loss is associated with reduced morbidity and mortality. The VA MOVE! program for weight loss is moderately effective but only reaches a small percentage of overweight Veterans. This proposed study will test whether a patient incentive program that gives Veterans non-financial incentives, such as Seattle Mariners baseball tickets, for losing one pound per week over 16 weeks is effective. An effective patient-incentive program could help more Veterans lose weight without requiring a substantial increase in VA staff.

DETAILED DESCRIPTION:
Project Background: Behavioral economics suggests that the chronic inability to make the daily behavioral changes that can help us lose weight may be the result of "present bias," which is a tendency to value small, immediate rewards over large rewards in the distant future. For many of us, the immediate gratification of eating an unhealthy food is a more powerful motivator than is the elusive dissatisfaction of the long-run health consequences of an unhealthy diet. Patient rewards may overcome present bias by moving the rewards for healthy behaviors forward in time. In a patient reward program, patients are given tangible, timely rewards for achieving specific health goals, such as losing one pound per week over 16 weeks. Meta analyses of randomized trials have found that rewards for weight loss are effective during the reward period, but the weight loss was not sustained after the reward was removed. Thus, the key challenge to a reward program is not achieving weight loss, but maintaining it. The proposed study tests the hypothesis that the significant weight regain found in prior reward trials can be attributed to use of financial rewards-e.g., cash or the equivalent of cash-in those trials. Experiments in behavioral economics have found that providing participants with financial rewards for participating in a study invokes behavior defined by reciprocity-the effort the participants gave in the study was proportional to the amount of money that they were given. When participants were given non-financial rewards, they exhibited no reciprocity-the effort was consistently high and did not vary with the quantity of the non-financial reward. By using financial rewards, prior trials may have invoked money-market norms of reciprocity, such that patients' efforts toward weight loss were high when rewards were offered, and reduced when they were discontinued. The investigators hypothesize that non-financial rewards, like tickets to a Seattle Mariners baseball game, will not invoke reciprocity or the consequent weight regain.

Project Objectives: The goal of this study is to test, through a randomized trial, the effectiveness of providing overweight Veterans with financial or non-financial rewards for a one pound weight loss per week over 16 weeks. The primary outcome is weight loss at 32 weeks-16 weeks after the discontinuation of the rewards. Secondary outcomes include weight loss at 16 weeks and 12 months.

Project Methods: The investigators will conduct a three-armed randomized trial of patient rewards for losing one pound per week over 16 weeks. The three treatment groups will receive financial rewards, non-financial rewards, or no rewards. The investigators hypothesize that: 1) patients who receive non-financial rewards for weight loss over 16 weeks will have greater weight loss at 32 weeks than patients who do not receive rewards; 2) patients who receive non-financial rewards for weight loss over 16 weeks will experience weight loss at 16 weeks that is not inferior to the weight loss of patients who receive financial rewards; and 3) weight regain will be greater among patients who received financial rewards compared to patients who received non-financial rewards or no rewards. The investigators will also conduct post-intervention qualitative interviews and perform a cost analysis.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* BMI>=30 at enrollment
* weigh less than 390lbs
* Active patient in primary care or women's clinic (1+ visit in last year)
* Access to a text capable phone in the Veteran's household or active email address
* live in Seattle area the entire year
* access to the internet

Exclusion Criteria:

* behavioral flag
* serious mental illness or anti-psychotic medication
* eating disorder and/or sexual trauma
* MOVE! participation in past 4 months
* pregnant or planning to become pregnant
* prisoner/employee/student
* inability to independently stand
* inability to read
* insulin dependent
* impaired decision making
* no access to a cell phone or phone that can receive text messages
* inability to remove socks & shoes
* >5% of body weight lost in last 6 months (clinical data and self-report)
* unable to pass cognitive screening

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul L. Hebert, PhD BA, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
A corresponding data repository has been created for this project. Participants must consent to both the main project and the data repository to be included in both. Otherwise the participant will only be included in this study.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 274 subjects consented to participate in the study, but 23 subjects did not complete the online baseline survey and did not respond to requests to complete the survey. Since randomization occurred after completion of the survey, only 251 subjects were randomized.
Groups:
- Financial Reward Arm: Financial rewards: Veterans in the financial reward arm receive all of the services of the usual care arm, plus rewards that are earned in two ways: an assured, and random. For the assured reward, they will receive compensation at the end of each month (defined as a four-week period) that they are at or below their target weight. For the random portion, each week that a participant is at or below their target weight, the patient is entered into a drawing to win additional compensation. Over the first eight weeks the patient has a 1-in-8 chance of winning. Over the 17-32-week period, Veterans in this group will receive token incentives for tracking and reporting their weekly weights regardless of whether it was on target. Each week that the patient enters their weight into the portal, they will have a 1-in-8 chance to earn the token incentive, such as a t-shirt or movie ticket. The participant will receive reminder text messages.
Period: Baseline to Week 16
Arm/Group | No Reward | Financial Reward Arm | Non-financial Reward Arm
Started | 73 | 91 | 87
Completed | 51 | 77 | 66
Not Completed | 22 | 14 | 21
Not completed — Lost to Follow-up | 8 | 10 | 16
Not completed — Withdrawal by Subject | 14 | 4 | 5
Period: Week 16 to 32
Arm/Group | No Reward | Financial Reward Arm | Non-financial Reward Arm
Started | 51 | 77 | 66
Completed | 40 | 67 | 60
Not Completed | 11 | 10 | 6
Not completed — Withdrawal by Subject | 3 | 3 | 1
Not completed — Lost to Follow-up | 8 | 7 | 5
Period: Week 32 to Week 52
Arm/Group | No Reward | Financial Reward Arm | Non-financial Reward Arm
Started | 40 | 67 | 60
Completed | 29 | 50 | 33
Not Completed | 11 | 17 | 27
Not completed — Lost to Follow-up | 11 | 16 | 27
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Reward | Financial Reward Arm | Non-financial Reward Arm | Total
Number analyzed (Participants) | 73 | 91 | 87 | 251
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (12.6) | 48.5 (12.6) | 49.6 (12.4) | 48.8 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 28 | 23 | 72
  Male | 52 | 63 | 64 | 179
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 20 | 3 | 33
  Not Hispanic or Latino | 63 | 71 | 84 | 218
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 15 | 9 | 17 | 41
  White | 43 | 70 | 52 | 165
  More than one race | 6 | 5 | 9 | 20
  Unknown or Not Reported | 6 | 6 | 4 | 16
Region of Enrollment [Number; unit: participants]
  United States | 73 | 91 | 87 | 251
Self Efficacy [Mean (Standard Deviation); unit: units on a scale] — Measured by survey responses to the Weight Efficacy Lifestyle Questionnaire Short Form (WEL-SF).Scale goes from 0 (not at all confident) to 10 (very confident). Higher scores mean better self efficacy.
  units on a scale | 6.6 (1.96) | 6.3 (2.20) | 6.3 (2.06) | 6.4 (2.08)
Intrinsic Motivation [Mean (Standard Deviation); unit: units on a scale] — Intrinsic motivation is measured by the Regulation of Eating Behaviors Scale. The score ranges for 1 to 7. Higher scores represent more intrinsic motivation to have a healthy diet.
  units on a scale | 4.0 (1.56) | 3.9 (1.58) | 4.4 (1.35) | 4.1 (1.52)
PHQ-8 Depression Score [Mean (Standard Deviation); unit: units on a scale] — Depression as measured by the PHQ-8. Scores range from 0 to 24. Higher scores represent more severe depression
  units on a scale | 10.5 (5.68) | 10.5 (5.56) | 10.4 (5.16) | 10.5 (5.44)

OUTCOME MEASURES:

1. Primary Outcome: Weight Change From Baseline to Week 32
Description: The primary outcome is weight measured in pounds at week 32 minus the weight at baseline.
Time Frame: 32 weeks
Population: Eligible Veterans at the VA Puget Sound Health Care Center who were age 18 to 69, had access to a text-capable mobile phone and had a BMI>=30. Exclusion criteria included conditions that affect the ability to participate in the trial (eating disorders, blindness, dementia, inability to read and weight>=390 lbs, which was the limit of the scales used); end-stage disease; pregnancy; and the use of antipsychotic medication.
Measure: Mean (97.5% Confidence Interval); unit: pounds
Groups:
- Control: At enrollment, participants randomized to usual care will be given the MOVE! workbook that serves both as an information resource on diet and exercise, a resource for tools to achieve weight loss goals, and a log of participants' goals, motivations, and outcomes. Each participant will be given a chart with a personalized target weight for a loss of 1lb. per week for 16 weeks. Participants will be given a digital scale or wireless scale and counseled to weigh themselves daily. Participants will enter their weight weekly into an online portal. They will also complete the surveys in the portal. They will receive text message reminders to enter their weight.
- Financial: Financial rewards: Veterans in the financial reward arm receive all of the services of the usual care arm, plus rewards that are earned in two ways: an assured, and random. For the assured reward, they will receive compensation at the end of each month (defined as a four-week period) that they are at or below their target weight. For the random portion, each week that a participant is at or below their target weight, the patient is entered into a drawing to win additional compensation. Over the first eight weeks the patient has a 1-in-8 chance of winning. Over the 17-32-week period, Veterans in this group will receive token incentives for tracking and reporting their weekly weights regardless of whether it was on target. Each week that the patient enters their weight into the portal, they will have a 1-in-8 chance to earn the token incentive, such as a t-shirt or movie ticket. The participant will receive reminder text messages.
- Non-Financial: Procedures for the non-financial rewards arm is identical to procedures for the financial reward arm, except that the Veteran will earn points rather than cash. Each week a random drawing will be for 20 points, each monthly weigh in is worth 5 points. Veterans will be given non-financial rewards associated with the number of points they earn.
Arm/Group | Control | Financial | Non-Financial
Number analyzed (Participants) | 40 | 67 | 60
pounds | -1.8 [-5.2 to 1.7] | -6.3 [-9.9 to 2.7] | -6.8 [-10.5 to -3.2]
Statistical Analysis 1: Comparison: Control vs Financial; Test type: Superiority; Mean Difference (Net) = -4.5, 97.5% CI 2-sided [-10.7 to 1.6] — Change in weight from baseline to week 32 in the financial rewards arm minus the change in weight from baseline to week 32 in the no rewards arm
Statistical Analysis 2: Comparison: Control vs Non-Financial; Test type: Superiority; p < 0.025, t-test, 2 sided; Mean Difference (Net) = -5.0, 97.5% CI 2-sided [-11.1 to 1] — Change in weight from baseline to week 32 in the non-financial arm minus the change in weight from baseline to week 32 in the no rewards arm

2. Secondary Outcome: Self Efficacy
Description: Measured by survey responses to the Weight Efficacy Lifestyle Questionnaire Short Form (WEL-SF).Scale goes from 0 (not at all confident) to 10 (very confident). Higher scores mean better outcomes. Missing values at follow-up were imputed using multiple imputation by chained equations (MICE)
Time Frame: Change form baseline to 16 weeks
Population: Two participants with missing data at baseline were dropped
Measure: Mean (97.5% Confidence Interval); unit: units on a scale
Arm/Group | No Reward | Financial Reward Arm | Non-financial Reward Arm
Number analyzed (Participants) | 73 | 90 | 86
units on a scale | -.7 [-1.5 to .1] | -.1 [-.8 to .6] | -.4 [-1.2 to .3]
Statistical Analysis 1: Comparison: No Reward vs Financial Reward Arm; Test type: Superiority; Mean Difference (Net) = 0.6, 97.5% CI 2-sided [-0.5 to 1.8] — Change in Self Efficacy score from baseline to week 16 in the financial rewards arm minus the change in Self Efficacy score from baseline to week 16 in the no rewards arm
Statistical Analysis 2: Comparison: No Reward vs Non-financial Reward Arm; Test type: Superiority; Mean Difference (Net) = 0.3, 97.5% CI 2-sided [-0.8 to 1.5] — Change in Self Efficacy score from baseline to week 16 in the nonfinancial rewards arm minus the change in Self Efficacy score from baseline to week 16 in the no rewards arm

3. Secondary Outcome: Self Efficacy
Description: Measured by survey responses to the Weight Efficacy Lifestyle Questionnaire Short Form (WEL-SF).Scale goes from 0 (not at all confident) to 10 (very confident).
Time Frame: Change form baseline to 32 weeks
Population: Missing values were imputed using multiple imputation by chained equations. Two participants were dropped for missing data at baseline survey.
Measure: Mean (97.5% Confidence Interval); unit: units on a scale
Arm/Group | No Reward | Financial Reward Arm | Non-financial Reward Arm
Number analyzed (Participants) | 73 | 90 | 86
units on a scale | -.4 [-1.4 to .6] | -.2 [-1.0 to 0.5] | .1 [-.7 to 0.9]
Statistical Analysis 1: Comparison: No Reward vs Financial Reward Arm; Test type: Superiority; Mean Difference (Net) = 0.1, 97.5% CI 2-sided [-1.2 to 1.4] — The change in self efficacy from baseline to week 32 in the financial incentive arm minus the change in self efficacy from baseline to week 32 in the no rewards arm
Statistical Analysis 2: Comparison: No Reward vs Non-financial Reward Arm; Test type: Superiority; Mean Difference (Net) = 0.5, 97.5% CI 2-sided [-.9 to 1.8] — The change in self efficacy from baseline to week 32 in the nonfinancial incentive arm minus the change in self efficacy from baseline to week 32 in the no rewards arm

4. Secondary Outcome: Self Efficacy
Description: as for outcome 3
Time Frame: Change form baseline to 52 weeks
Population: as for outcome 3
Measure: Mean (97.5% Confidence Interval); unit: units on a scale
Arm/Group | No Reward | Financial Reward Arm | Non-financial Reward Arm
Number analyzed (Participants) | 73 | 90 | 86
units on a scale | -1.4 [-2.5 to -0.4] | .1 [-.7 to .9] | -.3 [-1.1 to .5]
Statistical Analysis 1: Comparison: No Reward vs Financial Reward Arm; Test type: Superiority; Mean Difference (Net) = 1.5, 97.5% CI 2-sided [0.2 to 2.8] — The change in self efficacy from baseline to week 52 in the financial incentive arm minus the change in self efficacy from baseline to week 52 in the no rewards arm
Statistical Analysis 2: Comparison: No Reward vs Non-financial Reward Arm; Test type: Superiority; Mean Difference (Net) = 1.2, 97.5% CI 2-sided [0.0 to 2.3] — The change in self efficacy from baseline to week 52 in the nonfinancial incentive arm minus the change in self efficacy from baseline to week 52 in the no rewards arm

5. Secondary Outcome: Intrinsic Motivation
Description: Measured by patient survey responses to the Regulation of Eating Behavior Scale. Scale from 1 (does not agree at all) to 7 (agrees exactly). Higher values represent greater intrinsic motivation
Time Frame: Change form baseline to 16 weeks
Population: Two participants were dropped because of missing baseline data
Measure: Mean (97.5% Confidence Interval); unit: units on a scale
Arm/Group | No Reward | Financial Reward Arm | Non-financial Reward Arm
Number analyzed (Participants) | 73 | 90 | 86
units on a scale | -.4 [-.9 to .2] | -.1 [-.5 to .2] | -.3 [-.7 to 0.0]
Statistical Analysis 1: Comparison: No Reward vs Financial Reward Arm; Test type: Superiority; Mean Difference (Net) = 0.2, 97.5% CI 2-sided [-0.4 to 0.9] — Change in intrinsic motivation score from baseline to week 16 in the financial rewards arm minus the change in intrinsic motivation score from baseline to week 16 in the no rewards arm
Statistical Analysis 2: Comparison: No Reward vs Non-financial Reward Arm; Test type: Superiority; Mean Difference (Net) = 0.0, 97.5% CI 2-sided [-0.6 to 0.7] — Change in intrinsic motivation score from baseline to week 16 in the nonfinancial rewards arm minus the change in intrinsic motivation score from baseline to week 16 in the no rewards arm

6. Secondary Outcome: Intrinsic Motivation
Description: as for outcome 5
Time Frame: Change form baseline to 32 weeks
Population: as for outcome 3
Measure: Mean (97.5% Confidence Interval); unit: units on a scale
Arm/Group | No Reward | Financial Reward Arm | Non-financial Reward Arm
Number analyzed (Participants) | 73 | 90 | 86
units on a scale | -.7 [-1.3 to 0] | -.1 [-.7 to .4] | 0 [-.6 to .5]
Statistical Analysis 1: Comparison: No Reward vs Financial Reward Arm; Test type: Superiority; Mean Difference (Net) = 0.5, 97.5% CI 2-sided [-0.2 to 1.3] — The change in intrinsic motivation from baseline to week 32 in the financial incentive arm minus the change in intrinsic motivation from baseline to week 32 in the no rewards arm
Statistical Analysis 2: Comparison: No Reward vs Non-financial Reward Arm; Test type: Superiority; Mean Difference (Net) = 0.6, 97.5% CI 2-sided [-0.3 to 1.6] — The change in intrinsic motivation from baseline to week 32 in the nonfinancial incentive arm minus the change in intrinsic motivation from baseline to week 32 in the no rewards arm

7. Secondary Outcome: Intrinsic Motivation
Description: as for outcome 5
Time Frame: Change form baseline to 52 weeks
Population: as for outcome 3
Measure: Mean (97.5% Confidence Interval); unit: units on a scale
Arm/Group | No Reward | Financial Reward Arm | Non-financial Reward Arm
Number analyzed (Participants) | 73 | 90 | 86
units on a scale | -.6 [-1.6 to .4] | -.1 [-.7 to .5] | 0 [-.7 to .7]
Statistical Analysis 1: Comparison: No Reward vs Financial Reward Arm; Test type: Superiority; Mean Difference (Final Values) = 0.5, 97.5% CI 2-sided [-0.5 to 1.5] — The change in intrinsic motivation from baseline to week 52 in the financial incentive arm minus the change in intrinsic motivation from baseline to week 52 in the no rewards arm
Statistical Analysis 2: Comparison: No Reward vs Non-financial Reward Arm; Test type: Superiority; Mean Difference (Net) = 0.4, 97.5% CI 2-sided [-0.8 to 1.6] — Incentive Group minus usual care

8. Secondary Outcome: PHQ-8 Depression Score
Description: Measured by patient survey responses to the Personal Health Questionnaire Depression Scale (PHQ-8). The scale ranges from 0 to 24. Higher scores mean more severe depression.
Time Frame: Change from baseline to week 16
Population: Two subjects were dropped because they did not complete the baseline survey
Measure: Mean (97.5% Confidence Interval); unit: units on a scale
Arm/Group | No Reward | Financial Reward Arm | Non-financial Reward Arm
Number analyzed (Participants) | 73 | 90 | 86
units on a scale | -.2 [-2.2 to 1.9] | .1 [-1.1 to 1.3] | .6 [-0.7 to 1.8]
Statistical Analysis 1: Comparison: No Reward vs Financial Reward Arm; Test type: Superiority; Mean Difference (Net) = 0.3, 97.5% CI 2-sided [-2.0 to 2.6] — Change in PHQ-8 score from baseline to week 16 in the financial rewards arm minus the change in PHQ-8 score from baseline to week 16 in the no rewards arm
Statistical Analysis 2: Comparison: No Reward vs Non-financial Reward Arm; Test type: Superiority; Mean Difference (Net) = 0.7, 97.5% CI 2-sided [-1.5 to 2.9] — Change in PHQ-9 from week baseline to week 16 in the non-financial incentive group minus the change from week baseline to week 16 in the no rewards group

9. Secondary Outcome: PHQ-8 Depression Score
Description: Measured by patient survey responses to the Personal Health Questionnaire Depression Scale (PHQ-8). The scale has the following options: not at all, several days, more than half the days, nearly every day. Scores range from 0 to 24. Higher scores represent more severe depression.
Time Frame: change from baseline to 32 weeks
Population: as for outcome 3
Measure: Mean (97.5% Confidence Interval); unit: units on a scale
Arm/Group | No Reward | Financial Reward Arm | Non-financial Reward Arm
Number analyzed (Participants) | 73 | 90 | 86
units on a scale | -1.7 [-4.2 to .8] | -.3 [-2.1 to 1.5] | .5 [-1.4 to 2.4]
Statistical Analysis 1: Comparison: No Reward vs Financial Reward Arm; Test type: Superiority; Mean Difference (Net) = 1.4, 97.5% CI 2-sided [-1.7 to 4.5] — The change in PHQ-8 from baseline to week 32 in the financial incentive arm minus the change in PHQ-8 from baseline to week 32 in the no rewards arm
Statistical Analysis 2: Comparison: No Reward vs Non-financial Reward Arm; Test type: Superiority; Mean Difference (Net) = 2.2, 97.5% CI 2-sided [-0.7 to 5.0] — The change in PHQ-8 from baseline to week 32 in the nonfinancial incentive arm minus the change in PHQ-8 from baseline to week 32 in the no rewards arm

10. Secondary Outcome: PHQ-8 Depression Score
Description: Measured by patient survey responses to the Personal Health Questionnaire Depression Scale (PHQ-8). Measured by patient survey responses to the Personal Health Questionnaire Depression Scale (PHQ-8). The scale ranges from 0 to 24. Higher scores mean more severe depression.
Time Frame: change from baseline to 52 weeks
Population: as for outcome 3
Measure: Mean (97.5% Confidence Interval); unit: units on a scale
Arm/Group | No Reward | Financial Reward Arm | Non-financial Reward Arm
Number analyzed (Participants) | 73 | 90 | 86
units on a scale | .8 [-2.3 to 3.9] | -.3 [-2.3 to 1.8] | 1.1 [-0.9 to 3.1]
Statistical Analysis 1: Comparison: No Reward vs Financial Reward Arm; Test type: Superiority; Mean Difference (Net) = -1.1, 97.5% CI 2-sided [-4.9 to 2.8] — Change in PHQ-8 score from baseline to week 52 in the financial rewards arm minus the change in PHQ-8 score from baseline to week 52 in the no rewards arm
Statistical Analysis 2: Comparison: No Reward vs Non-financial Reward Arm; Test type: Superiority; Mean Difference (Net) = 0.3, 97.5% CI 2-sided [-2.9 to 3.6] — The change in PHQ-8 from baseline to week 52 in the nonfinancial incentive arm minus the change in PHQ-8 from baseline to week 52 in the no rewards arm

11. Secondary Outcome: Weight Change From Baseline
Description: A secondary outcome is weight measured in pounds at week 16 minus the weight at baseline.
Time Frame: 16 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: weight in pounds
Arm/Group | Control | Financial | Non-Financial
Number analyzed (Participants) | 51 | 77 | 66
weight in pounds | -2.4 [-5 to 0.3] | -5.6 [-8 to -3.1] | -7.0 [-9.4 to -4.5]
Statistical Analysis 1: Comparison: Control vs Financial; Test type: Superiority; Mean Difference (Net) = -3.2, 97.5% CI 2-sided [-7.4 to 1] — Change in weight from baseline to week 16 in the financial rewards arm minus the change in weight from baseline to week 16 in the no rewards arm
Statistical Analysis 2: Comparison: Control vs Non-Financial; Test type: Superiority; Mean Difference (Net) = -4.6, 97.5% CI 2-sided [-8.7 to -0.4] — Change in weight from baseline to week 16 in the nonfinancial rewards arm minus the change in weight from baseline to week 32 in the no rewards arm

12. Secondary Outcome: Weight Change From Baseline
Description: A secondary outcome is weight measured in pounds at week 52 minus the weight at baseline.
Time Frame: 52 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: weight in lbs
Arm/Group | Control | Financial | Non-Financial
Number analyzed (Participants) | 29 | 50 | 33
weight in lbs | -5.4 [-10.2 to 0.6] | -3 [-7.8 to 1.8] | -9 [-13.6 to 4.3]
Statistical Analysis 1: Comparison: Control vs Financial; Test type: Superiority; Mean Difference (Net) = 2.4, 97.5% CI 2-sided [-6 to 10.7] — Change in weight from baseline to week 52 in the financial rewards arm minus the change in weight from baseline to week 52 in the no rewards arm
Statistical Analysis 2: Comparison: Control vs Non-Financial; Test type: Superiority; Mean Difference (Net) = -3.6, 97.5% CI 2-sided [-11.2 to 4.1] — Change in weight from baseline to week 52 in the nonfinancial rewards arm minus the change in weight from baseline to week 52 in the no rewards arm

13. Other Pre Specified Outcome: Total Intervention Costs for All Participants
Description: The investigators will collect data on the cost of the intervention.
Time Frame: through 16 weeks
Population: All patients enrolled at baseline
Measure: Number; unit: dollars
Arm/Group | No Reward | Financial Reward Arm | Non-financial Reward Arm
Number analyzed (Participants) | 73 | 91 | 87
dollars | 0 | 21559 | 21754

ADVERSE EVENTS:
Time Frame: Up to 52 weeks.
Description: We used the clinicaltrials.gov definition.
Arm/Group | No Reward | Financial Reward Arm | Non-financial Reward Arm
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/91 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/91 | 0/87
Other Adverse Events (participants affected / at risk) | 0/73 | 0/91 | 0/87

LIMITATIONS AND CAVEATS:
The enrollment goal for the study was 280 participants. Enrollment and study recruitment was terminated on 3/4/2020 with 274 participants due to the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/39/NCT02957539/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-27): https://cdn.clinicaltrials.gov/large-docs/39/NCT02957539/ICF_001.pdf